CLINICAL TRIAL: NCT07084129
Title: Vancomycin and Acute Kidney Injury in Sepsis Treatment - Pharmacologic Modeling Intervention
Brief Title: Vancomycin and Acute Kidney Injury in Sepsis Treatment - Intervention
Acronym: VAST-i
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-022663; K23DK119463 (NIH)
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Sepsis
Keywords: sepsis; vancomycin; biomarker; pharmacokinetics
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Personalized vancomycin Pharmacokinetic model for dose adjustments (Experimental): Enrolled patients who are prescribed vancomycin by the clinical team will transition to the study-determined empiric vancomycin dosing at the time of enrollment, 12mg/kg/dose administered as an extended intravenous (IV) infusion over 2 hours given every 6 hours. Urinary neutrophil gelatinase-associated lipocalin (NGAL) will be measured as soon as possible after enrollment. Dosage adjustments will be made using the personalized vancomycin pharmacokinetic (PK) model incorporating the NGAL level once resulted. Daily urinary NGAL will be measured while on vancomycin therapy and in the intensive care unit (ICU) to evaluate for ongoing changes in renal function that may necessitate further dosage adjustments using the personalized vancomycin PK model, until clinically stabilized. Patients will undergo vancomycin area under the curve (AUC) monitoring with three timed blood draws for vancomycin concentrations with each vancomycin dosing change with a goal AUC target range of 400-600.
  Interventions: Other: personalized dosing adjustment of vancomycin

INTERVENTIONS:
Other: personalized dosing adjustment of vancomycin — A personalized vancomycin PK model that incorporates kidney injury biomarkers will be used for vancomycin dose adjustments to achieve goal AUC levels.

SUMMARY:
The goal of this clinical trial is to determine if vancomycin dosing in children with sepsis can be improved by using updated, personalized dosing models that account for new markers of an individual's kidney function. Vancomycin is prescribed based on the known information of how the body breaks this medicine down. Vancomycin may not be effective if blood levels of the medicine are too low. Vancomycin has potential side effects, including the possibility of injury to the kidney. These side effects usually happen when blood levels of vancomycin are too high. There are guidelines for the range of vancomycin blood levels doctors should target to treat an infection and lower the risk of side effects. Children with sepsis may metabolize vancomycin at different rates, faster or slower, than children who do not have sepsis. For these reasons, the current dosing strategy may lead to a higher risk of kidney injury or a risk of not adequately treating an infection in children with sepsis. The investigators' goal is to use new vancomycin dosing equations to improve the ability to select the right dose of vancomycin. The main questions this trial aims to answer are:

1. Is it feasible to use personalized models of vancomycin dosing in children with sepsis?
2. Will personalized models of vancomycin dosing achieve vancomycin blood levels in acceptable ranges?

ELIGIBILITY:
Inclusion Criteria:

1. Age >1 month and <18 years
2. Weight >5kg and <50kg
3. Vancomycin intended duration of therapy ≥48 hours
4. Admitted to intensive care unit with suspected or confirmed sepsis
5. Either sepsis-induced respiratory (invasive mechanical ventilation) or cardiovascular (vasoactive infusion) dysfunction as part of sepsis-associated organ dysfunction (these organ dysfunctions may be improving or resolved at the time of enrollment)

Exclusion Criteria:

1. Serum creatinine elevated and meets criteria for trough-based dosing by local Clinical Pharmacy
2. Methicillin resistant Staph aureus minimum inhibitory concentration (MIC)>1
3. Central nervous system infection
4. Extracorporeal support (extracorporeal membrane oxygenation, continuous renal replacement therapy)
5. Pregnancy
6. Patients on chronic dialysis therapy
7. Patients with known history of delayed vancomycin clearance based on local pharmacy records

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - personalized dose adjustment performed | From enrollment to the longer of 7 days after the completion of vancomycin therapy or through 30 days from enrollment
  Percentage of enrolled patients in which urinary neutrophil gelatinase-associated lipocalin is measured and used to make a vancomycin dosing recommendation

SECONDARY OUTCOMES:
Feasibility - Use of study-determined empiric vancomycin dosing | From enrollment to the longer of 7 days after the completion of vancomycin therapy or through 30 days from enrollment
  Percentage of patients transitioned to the study-determined empiric vancomycin dosing.
Feasibility - Area under the curve sampling attainment on study empiric vancomycin dosing | From study enrollment to the longer of 7 days after the completion of vancomycin therapy or through 30 days from enrollment
  Percentage of patients transitioned to the study-determined empiric vancomycin dosing and undergo subsequent area under the curve sampling.
Feasibility - Dosing change based on urinary neutrophil gelatinase-associated lipocalin level | From study enrollment to the longer of 7 days after the completion of vancomycin therapy or through 30 days from enrollment
  Percentage of patients enrolled in which urinary neutrophil gelatinase-associated lipocalin is used to make a dosing recommendation and results in administration of at least one adjusted dose of vancomycin.
Feasibility - Area under the curve sampling attainment after personalized dose adjustment | From study enrollment to the longer of 7 days after the completion of vancomycin therapy or through 30 days from enrollment
  Percentage of patients who undergo dose adjustment and have subsequent area under the curve sampling performed
Efficacy and safety - area under the curve in goal range | From study enrollment to the longer of 7 days after the completion of vancomycin therapy or through 30 days from enrollment
  Percentage of patients achieving area under the curve in goal range of 400-600mg-h/L.
Efficacy and safety - resolution of gram positive infection | From study enrollment to the longer of 7 days after the completion of vancomycin therapy or through 30 days from enrollment
  Percentage of patients with resolution of gram positive infection within the standard antibiotic duration for the infectious etiology.
Efficacy and safety - development of acute kidney injury | From study enrollment to the longer of 7 days after the completion of vancomycin therapy or through 30 days from enrollment
  Percentage of patients who develop acute kidney injury during the intervention.
Efficacy and safety - treatment failure | From study enrollment to the longer of 7 days after the completion of vancomycin therapy or through 30 days from enrollment
  Percentage of patients with treatment failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: De-identified IPD and supporting information will be shared upon request and review by the primary investigator. A data use agreement will need to be in place prior to sharing data.